CLINICAL TRIAL: NCT05024058
Title: A Multi-center, Randomized, Double-blind, Placebo Controlled Study to Investigate the Efficacy and Safety of Ligelizumab (QGE031) in the Treatment of Chronic Inducible Urticaria (CINDU) in Adolescents and Adults Inadequately Controlled With H1-antihistamines
Brief Title: Study of Efficacy and Safety of Ligelizumab in Adolescents and Adults With Chronic Inducible Urticaria Who Remain Symptomatic Despite Treatment With H1- Antihistamines
Acronym: PEARL-PROVOKE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Phase III PEARL studies (CQGE031C2302 and CQGE031C2303) with ligelizumab met their primary endpoint of superiority vs placebo at Week 12 for treatment of CSU, but not versus omalizumab. Decision to discontinue was not based on safety concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQGE031E12301; 2020-003018-11 (EudraCT Number)
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Chronic Inducible Urticaria
Keywords: ligelizumab; anti-IgE; CINDU; chronic inducible urticaria; symptomatic dermographism; cold urticaria; cholinergic urticaria; urticaria; itch; hives
MeSH Terms: conditions — Chronic Inducible Urticaria; Familial dermographism; Cold Urticaria; Urticaria; Pruritus | interventions — ligelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Ligelizumab low dose, symptomatic dermographism group (Experimental): Ligelizumab low dose subcutaneous injection every 4 weeks in participants with symptomatic dermographism
  Interventions: Drug: Ligelizumab
- Ligelizumab high dose, symptomatic dermographism (Experimental): Ligelizumab high dose subcutaneous injection every 4 weeks in participants with symptomatic dermographism
  Interventions: Drug: Ligelizumab
- Placebo SC q4W, symptomatic dermographism (Placebo Comparator): Placebo subcutaneous injection every 4 weeks in participants with symptomatic dermographism
  Interventions: Other: Placebo
- Ligelizumab low dose, cold urticaria (Experimental): Ligelizumab low dose subcutaneous injection every 4 weeks in participants with cold urticaria
  Interventions: Drug: Ligelizumab
- Ligelizumab high dose, cold urticaria (Experimental): Ligelizumab high dose subcutaneous injections every 4 weeks in participants with cold urticaria
  Interventions: Drug: Ligelizumab
- Placebo SC q4w, cold urticaria (Placebo Comparator): Placebo subcutaneous injection every 4 weeks in participants with cold urticaria
  Interventions: Other: Placebo
- Ligelizumab high dose, cholinergic urticaria (Experimental): Ligelizumab high dose subcutaneous injections every 4 weeks in participants with cholinergic urticaria
  Interventions: Drug: Ligelizumab
- Placebo SC q4w, cholinergic urticaria (Placebo Comparator): Placebo subcutaneous injections every 4 weeks in participants with cholinergic urticaria
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ligelizumab — Ligelizumab treated groups and arms
  Other Names: QGE031
  Arms: Ligelizumab high dose, cholinergic urticaria; Ligelizumab high dose, cold urticaria; Ligelizumab high dose, symptomatic dermographism; Ligelizumab low dose, cold urticaria; Ligelizumab low dose, symptomatic dermographism group
Other: Placebo — Placebo treated groups and arms
  Arms: Placebo SC q4W, symptomatic dermographism; Placebo SC q4w, cholinergic urticaria; Placebo SC q4w, cold urticaria

SUMMARY:
This was a placebo controlled, phase 3 study designed to evaluate the efficacy and safety of ligelizumab in participants with chronic inducible urticaria who are inadequately controlled with H1-antihistamines

DETAILED DESCRIPTION:
There are currently no approved therapies for patients with CINDU who remain symptomatic despite treatment with H1-antihistamines. The purpose of this study was to establish efficacy and safety of ligelizumab (QGE031) over placebo in participants with chronic inducible urticaria (CINDU) who remain symptomatic despite treatment with H1 antihistamine.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed CINDU diagnosis (as per guidelines) for symptomatic dermographism, cold urticaria or cholinergic urticaria for ≥ 4 months.

  * Diagnosis of CINDU (symptomatic dermographism, cold urticaria or cholinergic urticaria) inadequately controlled with H1-AH at local label approved doses at the time of randomization, as defined by all of the following:
  * Positive response (i.e development of symptoms) to triggers despite treatment with H1-AH
  * Positive response (i.e. development of symptoms) to provocation test on day of randomization
  * Participants must be able to physically perform the protocol defined provocation test specific to the participant's CINDU.
  * Cholinergic urticaria participants must show sweating in performing the pulse-controlled ergometry test on day of randomization. Participants with anhidrosis must not be included.
  * Willing and able to complete a daily symptom eDiary as per protocol requirement and adhere to the study visit schedules

Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or its components or to drugs of similar chemical classes or to the provocation test or items used in provocation tests

  * Participants who have concomitant CSU at screening
  * Participants who have a familial form of the target CINDU that is being considered for the participant's inclusion in this study
  * Participants having a more defined other form of inducible urticaria than the target CINDU that is being considered for the participant's inclusion in this study
  * Diseases, other than chronic inducible urticaria, with urticarial or angioedema symptoms such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary or acquired angioedema (eg, due to C1 inhibitor deficiency).
  * Any other skin disease associated with chronic itching that might influence, in the investigator's opinion, the study evaluations and results (eg, atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, etc.) or skin diseases associated with only wheals and no itch e.g asymptomatic dermographism
  * Prior exposure to ligelizumab, omalizumab and or other anti-IgE therapies

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (4):
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Murray, Utah
- Australia (2):
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Athens, Greece
- Hungary (3):
  - Novartis Investigative Site, Debrecen, Hajdú-Bihar
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Russia (4):
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
- Slovakia (2):
  - Novartis Investigative Site, Kežmarok
  - Novartis Investigative Site, Svidník
- Spain (3):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Taipei, Taiwan
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 participants were randomized. None completed study.
Pre-assignment Details: There were no pre-assignment details for this study.
Groups:
- 72 mg Ligelizumab, Symptomatic Dermographism: 72 mg ligelizumab subcutaneous injections every 4 weeks in participants with symptomatic dermographism
- 120 mg Ligelizumab, Symptomatic Dermographism: 120 mg ligelizumab subcutaneous injections every 4 weeks in participants with symptomatic dermographism
- Placebo - 72 mg Ligelizumab, Symptomatic Dermographism: Placebo every 4 weeks until week 12 followed by 72 mg ligelizumab subcutaneous injections in participants with symptomatic dermographism
- Placebo - 120 mg Ligelizumab, Symptomatic Dermographism: Placebo every 4 weeks until week 12 followed by 120 mg ligelizumab subcutaneous injections in participants with symptomatic dermographism
- 72 mg Ligelizumab Cold Urticaria: 72 mg ligelizumab subcutaneous injections every 4 weeks in participants with cold urticaria
- 120 mg Ligelizumab, Cold Urticaria: 120 mg ligelizumab subcutaneous injections every 4 weeks in participants with cold urticaria
- Placebo - 72 mg Ligelizumab, Cold Urticaria: Placebo every 4 weeks until week 12 followed by 72 mg ligelizumab subcutaneous injections in participants with cold urticaria
- Placebo - 120 mg Ligelizumab, Cold Urticaria: Placebo every 4 weeks until week 12 followed by 120 mg ligelizumab subcutaneous injections in participants with cold urticaria
- 120 mg Ligelizumab, Cholinergic Urticaria: 120 mg ligelizumab subcutaneous injection every 4 weeks in participants with cholinergic urticaria
- Placebo - 120 mg Ligelizumab, Cholinergic Urticaria: Placebo every 4 weeks until week 12 followed by 120 mg ligelizumab subcutaneous injections in participants with cholinergic urticaria
Period: Treatment
Arm/Group | 72 mg Ligelizumab, Symptomatic Dermographism | 120 mg Ligelizumab, Symptomatic Dermographism | Placebo - 72 mg Ligelizumab, Symptomatic Dermographism | Placebo - 120 mg Ligelizumab, Symptomatic Dermographism | 72 mg Ligelizumab Cold Urticaria | 120 mg Ligelizumab, Cold Urticaria | Placebo - 72 mg Ligelizumab, Cold Urticaria | Placebo - 120 mg Ligelizumab, Cold Urticaria | 120 mg Ligelizumab, Cholinergic Urticaria | Placebo - 120 mg Ligelizumab, Cholinergic Urticaria
Started | 5 | 6 | 4 | 2 | 3 | 3 | 1 | 3 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 6 | 4 | 2 | 3 | 3 | 1 | 3 | 6 | 6
Not completed — Study terminated by sponsor | 5 | 6 | 4 | 2 | 3 | 3 | 1 | 3 | 6 | 6
Period: Follow-up
Arm/Group | 72 mg Ligelizumab, Symptomatic Dermographism | 120 mg Ligelizumab, Symptomatic Dermographism | Placebo - 72 mg Ligelizumab, Symptomatic Dermographism | Placebo - 120 mg Ligelizumab, Symptomatic Dermographism | 72 mg Ligelizumab Cold Urticaria | 120 mg Ligelizumab, Cold Urticaria | Placebo - 72 mg Ligelizumab, Cold Urticaria | Placebo - 120 mg Ligelizumab, Cold Urticaria | 120 mg Ligelizumab, Cholinergic Urticaria | Placebo - 120 mg Ligelizumab, Cholinergic Urticaria
Started | 2 | 5 | 4 | 0 | 3 | 2 | 0 | 2 | 5 | 6
Completed | 1 | 5 | 3 | 0 | 3 | 2 | 0 | 1 | 5 | 5
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Randomized Analysis Set (RAN) consisted of all randomized participants, regardless of whether or not they received a dose of study drug. Participants were analyzed according to the treatment they were assigned. Data could not be analyzed because no subject completed Week 12 in the sympomatic dermographism cohort, 1 subject each completed the Week 12 in 72 mg ligelizumab and 120 mg ligelizumab groups in cold urticaria cohort, 1 subject completed Week 12 in cholinergic urticaria cohort.
Groups:
- Placebo - 120 mg Ligelizumab, Cold Urticaria: Placebo every 4 weeks until week 12 followed by 72 mg ligelizumab subcutaneous injections in participants with cold urticaria
- Total: Total of all reporting groups
Arm/Group | 72 mg Ligelizumab, Symptomatic Dermographism | 120 mg Ligelizumab, Symptomatic Dermographism | Placebo - 72 mg Ligelizumab, Symptomatic Dermographism | Placebo - 120 mg Ligelizumab, Symptomatic Dermographism | 72 mg Ligelizumab Cold Urticaria | 120 mg Ligelizumab, Cold Urticaria | Placebo - 72 mg Ligelizumab, Cold Urticaria | Placebo - 120 mg Ligelizumab, Cold Urticaria | 120 mg Ligelizumab, Cholinergic Urticaria | Placebo - 120 mg Ligelizumab, Cholinergic Urticaria | Total
Number analyzed (Participants) | 5 | 6 | 4 | 2 | 3 | 3 | 1 | 3 | 6 | 6 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 5
  Between 18 and 65 years | 4 | 5 | 3 | 2 | 3 | 2 | 1 | 2 | 6 | 6 | 34
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (9.81) | 28.3 (12.74) | 40.8 (18.86) | 36.5 (12.02) | 35.3 (12.50) | 31.7 (16.17) | 60.0 (NA) — Not evaluable | 32.3 (26.58) | 28.8 (9.62) | 25.2 (5.56) | 27.0 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 2 | 3 | 2 | 1 | 1 | 2 | 0 | 19
  Male | 2 | 3 | 2 | 0 | 0 | 1 | 0 | 2 | 4 | 6 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 6 | 4 | 2 | 3 | 3 | 1 | 3 | 5 | 5 | 36
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Fric Score in Participants With Symptomatic Dermographism
Description: Total Fric score (a scale of 0-4 where 0= no linear hive ≥ 3mm in width, 1= one linear hive ≥ 3mm in width, 2= two linear hives ≥ 3mm in width, 3= three linear hives ≥ 3mm in width and 4 = four linear hives ≥ 3mm in width)
  None of the participants completed Week 12 and hence at Week 12 was not analyzed
Time Frame: Baseline, Week 12
Population: The Randomized Analysis Set (RAN) consisted of all randomized participants, regardless of whether or not they received a dose of drug. Participants were analyzed according to the treatment they were assigned.
  Due to the limited number of participants who completed the primary endpoint timepoint (Week 12), no inferential statistical analysis was done for primary and secondary endpoints.
Groups:
- 72 mg Ligelizumab, Symptomatic Dermographism: 72 mg ligelizumab subcutaneous injection every 4 weeks in participants with symptomatic dermographism
- Placebo -120 mg Ligelizumab, Symptomatic Dermographism: Placebo every 4 weeks until week 12 followed by 120 mg ligelizumab subcutaneous injections in participants with symptomatic dermographism
Arm/Group | 72 mg Ligelizumab, Symptomatic Dermographism | 120 mg Ligelizumab, Symptomatic Dermographism | Placebo - 72 mg Ligelizumab, Symptomatic Dermographism | Placebo -120 mg Ligelizumab, Symptomatic Dermographism
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Critical Temperature Threshold in Participants With Cold Urticaria
Description: The TempTest is used to induce itch and hives in participants with cold urticaria. Critical temperature threshold (CTT), as measured by the TempTest, determines the highest temperature sufficient for inducing symptoms.
Time Frame: Baseline, Week 12
Population: RAN consisted of all randomized participants, regardless of whether or not they received a dose of drug. Participants were analyzed according to the treatment they were assigned.
  Due to the limited number of participants who completed the primary endpoint timepoint (Week 12), no inferential statistical analysis was done for primary and secondary endpoints.
Measure: Number; unit: Temperature (degrees celcius)
Groups:
- 72 mg Ligelizumab Cold Urticaria: 72 mg ligelizumab subcutaneous injection every 4 weeks in participants with cold urticaria
Arm/Group | 72 mg Ligelizumab Cold Urticaria | 120 mg Ligelizumab, Cold Urticaria | Placebo - 72 mg Ligelizumab, Cold Urticaria | Placebo - 120 mg Ligelizumab, Cold Urticaria
Number analyzed (Participants) | 1 | 1 | 0 | 0
Temperature (degrees celcius) | -26 | -15 |  |

3. Primary Outcome: Change From Baseline in Itch Numerical Rating Scale in Participants With Cholinergic Urticaria
Description: Itch numerical rating scale, a scale from 0 to 10. Negative change from baseline indicates improvement.
  Patients were asked to rate itching severity based on the worst level of itching in the past 24 h using an 11-point scale from 0 ("no itch") to 10 ("worst possible itch")
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Number; unit: Scores on a scale
Groups:
- 120 mg Ligelizumab, Cholinergic Urticaria: 120 mg ligelizumab subcutaneous injections in participants with cholinergic urticaria
Arm/Group | 120 mg Ligelizumab, Cholinergic Urticaria | Placebo - 120 mg Ligelizumab, Cholinergic Urticaria
Number analyzed (Participants) | 1 | 0
Scores on a scale | -7 |

4. Secondary Outcome: Proportion of Participants With Symptomatic Dermographism With Total Fric Score = 0
Description: Total Fric score (a scale of 0-4 where 0= no linear hive ≥ 3mm in width, 1= one linear hive ≥ 3mm in width, 2= two linear hives ≥ 3mm in width, 3= three linear hives ≥ 3mm in width and 4 = four linear hives ≥ 3mm in width)
  None of the participants completed Week 12
Time Frame: Week 12
Population: as for outcome 2
Arm/Group | 72 mg Ligelizumab, Symptomatic Dermographism | 120 mg Ligelizumab, Symptomatic Dermographism | Placebo - 72 mg Ligelizumab, Symptomatic Dermographism | Placebo - 120 mg Ligelizumab, Symptomatic Dermographism
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Itch Numerical Rating Scale in Participants With Symptomatic Dermographism
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: RAN consisted of all randomized participants, regardless of whether or not they received a dose of drug. Participants were analyzed according to the treatment they were assigned.
  No participants completed week 12.
Arm/Group | 72 mg Ligelizumab, Symptomatic Dermographism | 120 mg Ligelizumab, Symptomatic Dermographism | Placebo - 72 mg Ligelizumab, Symptomatic Dermographism | Placebo - 120 mg Ligelizumab, Symptomatic Dermographism
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Proportion of Participants With Cold Urticaria With Complete Response (no Itch or Hives) to the TempTest
Description: The TempTest® is used to induce itch and hives in participants with cold urticaria. Critical temperature threshold (CTT), as measured by the TempTest, determines the highest temperature sufficient for inducing symptoms.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Number; unit: Proportion of participants
Groups:
- 72 mg Ligelizumab, Cold Urticaria: 72 mg ligelizumab subcutaneous injections every 4 weeks in participants with cold urticaria
Arm/Group | 72 mg Ligelizumab, Cold Urticaria | 120 mg Ligelizumab, Cold Urticaria | Placebo - 72 mg Ligelizumab, Cold Urticaria | Placebo - 120 mg Ligelizumab, Cold Urticaria
Number analyzed (Participants) | 1 | 1 | 0 | 0
Proportion of participants | 1 | 0 |  |

7. Secondary Outcome: Change From Baseline in Itch Numerical Rating Scale in Participants With Cold Urticaria
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Number; unit: Scores on a scale
Groups:
- Placebo - 72 mg Ligelizumab, Cold Urticaria: Placebo every 4 weeks until week 12 followed by 72 mg ligelizumab subcutaneous injections in participants with symptomatic dermographism
- Placebo -120 mg Ligelizumab, Cold Urticaria: Placebo every 4 weeks until week 12 followed by 72 mg ligelizumab subcutaneous injections in participants with cold urticaria
Arm/Group | 72 mg Ligelizumab Cold Urticaria | 120 mg Ligelizumab, Cold Urticaria | Placebo - 72 mg Ligelizumab, Cold Urticaria | Placebo -120 mg Ligelizumab, Cold Urticaria
Number analyzed (Participants) | 1 | 1 | 0 | 0
Scores on a scale | -9 | 0 |  |

8. Secondary Outcome: Proportion of Participants With Cholinergic Urticaria With Itch Numerical Rating Scale =0
Description: as for outcome 3
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Proportion of participants
Arm/Group | 120 mg Ligelizumab, Cholinergic Urticaria | Placebo - 120 mg Ligelizumab, Cholinergic Urticaria
Number analyzed (Participants) | 1 | 1
Proportion of participants | 0 | 0

9. Secondary Outcome: Proportion of Participants With Cholinergic Urticaria With Physician Global Assessment of Severity of Hives (PGA - Hive Score) =0
Description: Physician global assessment of severity of hives
  PGA is an assessment of all lesions scored on a scale from 0-5 (with 0 = No hives and 5 = Very severe hives)
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Proportion of participants
Arm/Group | 120 mg Ligelizumab, Cholinergic Urticaria | Placebo - 120 mg Ligelizumab, Cholinergic Urticaria
Number analyzed (Participants) | 1 | 0
Proportion of participants | 0 |

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected after signature of the informed consent form until 16 weeks from last dose (12 weeks from end of treatment). Treatment period was 24 weeks. Serious Adverse Events (SAEs) were collected after signature of the informed consent form until 16 weeks from last dose (12 weeks from end of treatment).
Description: AEs are any sign or symptom that occurs during conduct of trial and safety follow-up. AEs were reported per intervention and not combined. All AEs reported during Placebo-Ligelizumab 72mg and Placebo-Ligelizumab 120 mg occurred in placebo duration.
Groups:
- Ligelizumab 72mg: 72 mg ligelizumab subcutaneous injection every 4 weeks in participants with symptomatic dermographism
- Ligelizumab 120mg: symptomatic dermographism 120 mg ligelizumab subcutaneous injections every 4 weeks in participants with symptomatic
- Placebo - Ligelizumab 72mg: symptomatic dermographism Placebo every 4 weeks until week 12 followed by 72 mg ligelizumab subcutaneous injections in participants with symptomatic dermographism
- Placebo - Ligelizumab 120mg: symptomatic dermographism Placebo every 4 weeks until week 12 followed by 120 mg ligelizumab subcutaneous injections in participants with symptomatic dermographism
- Total: Total number of participants who participated in the trial
Arm/Group | Ligelizumab 72mg | Ligelizumab 120mg | Placebo - Ligelizumab 72mg | Placebo - Ligelizumab 120mg | Total
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/15 | 0/5 | 0/11 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/15 | 0/5 | 0/11 | 0/39
Other Adverse Events (participants affected / at risk) | 3/8 | 6/15 | 3/5 | 1/11 | 13/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ligelizumab 72mg (N=8) | Ligelizumab 120mg (N=15) | Placebo - Ligelizumab 72mg (N=5) | Placebo - Ligelizumab 120mg (N=11) | Total (N=39)
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 2
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT05024058/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT05024058/SAP_001.pdf